CLINICAL TRIAL: NCT02054650
Title: Osteopathic Manipulative Treatment of Somatic Dysfunction and Chronic Low Back Pain in Patients With Type 2 Diabetes Mellitus
Brief Title: OMT of Somatic Dysfunction and Chronic Low Back Pain in Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Scheduling and recruitment difficulties
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: American Osteopathic Association (Other); Osteopathic Heritage Foundations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-127; 13-11-686 (Other Grant/Funding Number: American Osteopathic Association)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Low Back Pain; Type 2 Diabetes Mellitus
Keywords: Chronic low back pain; Type 2 diabetes mellitus; Back pain; Diabetes; Osteopathic manual treatment; Osteopathic manipulative treatment; OMT; Biomarkers; Glycemic control; Kidney function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Back Pain; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osteopathic Manual Treatment (OMT) (Experimental): The OMT protocol will be delivered following an examination for somatic dysfunction at each treatment session. The protocol will target the thoracic, lumbosacral, iliac, and pubic regions using the following techniques: high-velocity, low-amplitude thrusts; moderate-velocity, moderate-amplitude thrusts; soft tissue including stretching, kneading, and pressure; myofascial stretching and release; counterstrain; muscle energy; and other optional techniques as time permits and indicated. The intervention will be delivered at weeks 0, 1, 2, 4, 6 and 8. Week 12 is a data collection visit with no intervention.
  Interventions: Other: Osteopathic Manual Treatment (OMT)
- Sham OMT (Sham Comparator): Sham OMT will involve hand contact, active and passive range of motion, and sham techniques that simulate OMT (including optional OMT techniques), but that utilize such maneuvers as light touch, improper patient positioning, purposely misdirected movements, and diminished provider force. Sham OMT will be delivered at weeks 0, 1, 2, 4, 6 and 8. Week 12 is a data collection visit with no intervention.
  Interventions: Other: Sham OMT

INTERVENTIONS:
Other: Osteopathic Manual Treatment (OMT) — Osteopathic Manual Treatment (OMT) is a system of hands-on techniques used by osteopathic physicians to increase function and reduce pain.
  Arms: Osteopathic Manual Treatment (OMT)
Other: Sham OMT — Sham OMT involves hand contact, active and passive range of motion, and sham techniques that simulate OMT, but that utilize such maneuvers as light touch, improper patient positioning, purposely misdirected movements, and diminished provider force.
  Arms: Sham OMT

SUMMARY:
The study hypothesis is based on osteopathic medical philosophy that: 1) the body is a unit; 2) the body has inherent self-regulatory mechanisms; 3) structure and function are interrelated; and 4) rational treatment is based on an understanding and integration of these concepts. Patients with type 2 diabetes mellitus often report more aches and pains than people without diabetes. Because osteopathic manual medicine addresses dysfunction in the musculoskeletal system, patients with both chronic low back pain and type 2 diabetes mellitus may benefit from this non-pharmacological treatment to reduce their pain, thereby reducing their stress and perhaps providing better clinical control for diabetes as demonstrated by key markers such as hemoglobin A1c and kidney function. This study is an extension of research completed in the OSTEOPATHIC Trial. Results of that study were published in the Annals of Family Medicine in March/April 2013.

DETAILED DESCRIPTION:
SPECIFIC AIM 1:

To conduct a randomized controlled trial (RCT) to determine the efficacy of osteopathic manual treatment (OMT) vs sham OMT in subjects with type 2 diabetes mellitus (T2DM) and comorbid chronic low back pain (LBP). This will involve a 12-week protocol to study changes in response to OMT in such outcomes as LBP severity (primary outcome measure), somatic dysfunction, renal function, glycemic control, and other biomarkers potentially related to T2DM.

SPECIFIC AIM 2:

Within the RCT, to corroborate previous findings indicating that patients with T2DM have a high prevalence of tissue texture abnormalities in the T11-L2 spinal segmental region and to determine if such findings can be statistically associated with the presence of diabetic nephropathy using such laboratory measures as serum creatinine, urinary microalbuminuria and macroalbuminuria, and the glomerular filtration rate.

SPECIFIC AIM 3:

Within the RCT, to explore potential mechanisms of action of OMT by longitudinally measuring concentrations of biomarkers such as insulin, glucagon, cortisol, hemoglobin A1c, tumor necrosis factor-α,interleukin (IL)-1β, IL-6, IL-10, and IL-18 in subjects with T2DM and comorbid chronic LBP over 12 weeks. Significant changes in biomarker concentrations may help explain the effects of OMT and whether such effects are mediated by changes in somatic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting plasma glucose ≥126 mg/dL; OR
2. Oral glucose tolerance test ≥200 mg/dL; OR
3. HbA1c ≥6.5%

   AND
4. Low back pain on most days for past three months; AND
5. Usual low back pain severity of 4 or greater on an 11 point numerical scale during the past week.

Exclusion Criteria:

1. age less than 18 years or age greater than 79 years; OR
2. having a previous or current diagnosis of type 1 diabetes mellitus; OR
3. having a history of any of the following pancreatic or related disorders: (a) acute or chronic pancreatitis, (b) pancreatic tumor or cancer, (c) Zollinger-Ellison syndrome, or (d) any other medical or surgical condition resulting in functional hypo- or hyperglycemia; OR
4. having end-stage renal disease; OR
5. having a history of any surgery involving the pancreas; OR
6. having a history of low back surgery in the past year; OR
7. receiving workers' compensation benefits in the past three months; OR
8. having involvement in ongoing litigation relating to diabetes mellitus or back problems; OR
9. having a history of a stroke or transient ischemic attack in the past year; OR
10. having used intravenous, intramuscular or oral corticosteroids within the past month; OR
11. attending a manual treatment session (OMT or any manual therapies delivered by chiropractors or physical therapists) in the past three months, or more than three times in the past year; OR
12. practicing osteopathic medicine, chiropractic, or physical therapy, or attending a corresponding professional school; OR
13. being pregnant; OR
14. currently participating in another medical research study

Subjects will also be excluded if any of the following conditions are found during the clinical screening:

1. presence of "red flag" conditions relating to LBP (cancer at any anatomical site, spinal osteomyelitis, spinal fracture, herniated disc, ankylosing spondylitis, or cauda equina syndrome); OR
2. angina or congestive heart failure symptoms with minimal activity; OR
3. active bleeding or infection in the lower back, or any other condition that might impede protocol implementation; OR
4. discovery of the presence of any telephone screening exclusion criterion (EXCEPT that the usual LBP severity over the past week may have declined from ≥4/10 points to ≥3/10 points during the lag time between screenings).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in low back pain severity | 12 weeks
  The change in low back pain severity will be measured using an 11-point numerical scale (0 to 10). The baseline measurement for each subject will be compared with the week 12 measurement to determine if a reduction in pain has occurred.

SECONDARY OUTCOMES:
Change in back-specific functioning | 12 weeks
  The change in back-specific functioning will be measured using the Roland-Morris Disability Questionnaire (scored from 0 to 24). The baseline measurement for each subject will be compared with the week 12 measurement to determine if an improvement in back-specific functioning has occurred.
Change in general health | 12 weeks
  The change in general health will be measured using the Short Form 36 Health Status Survey (scored from 0 to 100). The baseline measurement for each subject will be compared with the week 12 measurement to determine if an improvement in general health has occurred.
Change in glycemic control | 12 weeks
  The change in glycemic control will be measured using hemoglobin A1C levels. The baseline measurement for each subject will be compared with the week 12 measurement to determine if an improvement in glycemic control has occurred.
Tissue texture changes | 12 weeks
  The change in tissue texture will be assessed during physical examinations. The baseline findings for each subject will be compared with the week 12 findings to determine if a change in tissue texture has occurred.
Change in biomarker concentrations | 12 weeks
  Concentrations of biomarkers such as insulin, glucagon, cortisol, TNF-α, IL-1β, IL-6, IL-10, and IL-18 will be measured at baseline and at week 12 to determine if any significant change in a biomarker has occurred.

CONTACTS AND LOCATIONS:
Overall Officials: John C. Licciardone, DO, MS, MBA, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Licciardone JC, Kearns CM, Hodge LM, Minotti DE. Osteopathic manual treatment in patients with diabetes mellitus and comorbid chronic low back pain: subgroup results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2013 Jun;113(6):468-78. PMID 23739758
- [Background] Licciardone JC, Kearns CM, Minotti DE. Outcomes of osteopathic manual treatment for chronic low back pain according to baseline pain severity: results from the OSTEOPATHIC Trial. Man Ther. 2013 Dec;18(6):533-40. doi: 10.1016/j.math.2013.05.006. Epub 2013 Jun 10. PMID 23759340
- [Background] Licciardone JC, Minotti DE, Gatchel RJ, Kearns CM, Singh KP. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: a randomized controlled trial. Ann Fam Med. 2013 Mar-Apr;11(2):122-9. doi: 10.1370/afm.1468. PMID 23508598
- [Background] Licciardone JC, Kearns CM, Hodge LM, Bergamini MV. Associations of cytokine concentrations with key osteopathic lesions and clinical outcomes in patients with nonspecific chronic low back pain: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Sep;112(9):596-605. doi: 10.7556/jaoa.2012.112.9.596. PMID 22984233
- [Background] Licciardone JC, Kearns CM. Somatic dysfunction and its association with chronic low back pain, back-specific functioning, and general health: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Jul;112(7):420-8. PMID 22802542
- [Background] Licciardone JC, Gatchel RJ, Kearns CM, Minotti DE. Depression, somatization, and somatic dysfunction in patients with nonspecific chronic low back pain: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Dec;112(12):783-91. PMID 23212429
- [Background] Licciardone JC, Fulda KG, Stoll ST, Gamber RG, Cage AC. A case-control study of osteopathic palpatory findings in type 2 diabetes mellitus. Osteopath Med Prim Care. 2007 Feb 8;1:6. doi: 10.1186/1750-4732-1-6. PMID 17371582